CLINICAL TRIAL: NCT05770752
Title: Effect of Mechanical Ventilation on Peripheral Lymphatic Function - do Elevated Intrathoracic Pressure Impact Lymphatic Flow?
Brief Title: Lymphatic Function During Mechanical Ventilation
Acronym: LYMPH-UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lene Thorup, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P-2022-462
Record Dates: First submitted 2023-01-25; First posted 2023-03-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lymphatic Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Elevated pressure ventilation — Elevated pressure ventilation is defined as a raise in PIP and PEEP by 10 cmH2O from each patients original pressure setting, although never higher than a PIP of 30 cmH2O.

SUMMARY:
This study wil examine the effect of altered intrathoracic pressure on lymphatic function, by investigating the lymphatic vessels in the lower limb during mechanical ventilation.

The lymphatic function will be examined using Near-Infrared Fluorescence Imaging.

DETAILED DESCRIPTION:
This study wil examine the effect of altered intrathoracic pressure on lymphatic function. This will be done by investigating peripheral lymphatic vessels on patients undergoing surgery for malformations of the jaw who are being mechanically ventilated.

Subjects will be examined on two occasions. One to establish baseline function, and one during surgery following a ventilation protocol with altered PIP and PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for jaw malformations
* Age > 18 years
* Informed consent
* Cardiopulmonary healthy

Exclusion Criteria:

* History of Cardiac disease
* History of pulmonary disease
* History of lymphatic disease
* Peripheral edema
* Chronic infectious disease
* Age > 30 years
* BMI > 30

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Peripheral lymphatic velocity (centimeters/second) | 3 hours
  Peripheral lymphatic fluid velocity (centimeters/second) will be calculated based upon NIRF sequences.
Peripheral lymphatic frequency (contractions/minute) | 3 hours
  Peripheral lymphatic contraction frequency (contractions/minute) will be calculated based upon NIRF sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thorup, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark